CLINICAL TRIAL: NCT05686889
Title: Post-Hoc Enthusiasm and Wariness
Acronym: PHEW
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Don Redelmeier, Senior Scientist, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 5692
Record Dates: First submitted 2023-01-07; First posted 2023-01-17 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Health Behavior
MeSH Terms: conditions — Health Behavior | interventions — Self Report

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Success (Experimental): Symptomatic improvement present
  Interventions: Other: Patient self-report
- Failure (Experimental): Symptomatic improvement absent
  Interventions: Other: Patient self-report

INTERVENTIONS:
Other: Patient self-report — Simulated patient following structured script

SUMMARY:
The post-hoc fallacy (also termed the post-hoc-ergo-propter-hoc fallacy) has been recognized for centuries with endless relevance. The general concept in medical care is that patients who improve after a treatment are not necessary patients who improve because of a treatment. Modern medicine provides multiple opportunities to examine such pitfalls of judgment due to the prevailing uncertainty, incompleteness of our understanding pathogenic mechanisms, and natural tendency to connect treatments to outcomes. In this study, we will investigate whether judgments about vitamin supplementation might demonstrate the post-hoc fallacy.

DETAILED DESCRIPTION:
We plan to conduct a brief survey of pharmacies portraying a patient in two slightly different versions. One version will portray the patient who feels better after starting a vitamin supplement whereas another version will portray the patient who feels unchanged after starting a vitamin supplement. The patients will be randomly assigned to participants and otherwise contain identical information. Judgments will be measured by eliciting participants recommendation about continuing the vitamin (Appendix_Script).

ELIGIBILITY:
Inclusion Criteria:

* Community pharmacist

Exclusion Criteria:

* Outside Ontario

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Response variable in each survey is a binary recommendation whether to continue the vitamin supplement or discontinue the vitamin supplement | Short-term (less than 5 minutes)
  Health provider clinical recommendation

CONTACTS AND LOCATIONS:
Overall Officials: Donald A Redelmeier, MD, MSc, Principal Investigator — Sunnybrook Health Sciences Centre

IPD SHARING:
Plan to Share IPD: No